CLINICAL TRIAL: NCT06389279
Title: The Effect of Ultrasound-guided Pericapsular Nerve Block, Fascia Iliaca Compartment Block and Femoral Block on Postoperative Recovery Quality in Hip Surgery
Brief Title: The Effect of Facial Plane Blocks on Postoperative Recovery Quality in Hip Surgery
Status: Recruiting | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-18/11
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hip Fracture
Keywords: regional anesthesia; postoperative pain; recovery quality; hip fracture
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PENG block group: Before the spinal anesthesia, PENG block will be performed under the guidance of ultrasound.
  Interventions: Other: PENG block group
- FIC block group: Before the spinal anesthesia, FIC block will be performed under the guidance of ultrasound.
  Interventions: Other: FIC block group
- Femoral block group: Before the spinal anesthesia, femoral block will be performed under the guidance of ultrasound.
  Interventions: Other: Femoral block group
- Control group: No intervention
  Interventions: Other: Control group

INTERVENTIONS:
Other: PENG block group — Ultrasound-guided PENG block is performed approximately 30 minutes before surgery in patients undergoing hip surgery in a separate regional anaesthesia room with standard anaesthesia monitoring.
  Groups: PENG block group
Other: FIC block group — Ultrasound-guided FIC block is performed approximately 30 minutes before surgery in patients undergoing hip surgery in a separate regional anaesthesia room with standard anaesthesia monitoring.
  Groups: FIC block group
Other: Femoral block group — Ultrasound-guided femoral block is performed approximately 30 minutes before surgery in patients undergoing hip surgery in a separate regional anaesthesia room with standard anaesthesia monitoring.
  Groups: Femoral block group
Other: Control group — No intervention
  Groups: Control group

SUMMARY:
The aim of this study was to evaluate the effect of ultrasound-guided pericapsular nerve block, fascia iliaca compartment block, and femoral block on the quality of recovery as part of multimodal analgesia before hip surgery under spinal anesthesia.

DETAILED DESCRIPTION:
Orthopedic procedures have become increasingly common in clinical practice. With the increasing elderly population, there have been significant developments in recent years in the field of perioperative pain management and anesthesia strategies for patients scheduled for hip surgery. Patients undergoing hip surgery may experience severe pain both postoperatively and during the positioning of the patient during surgery. This leads to increased sympathetic activation such as tachycardia and hypertension in patients, especially in the elderly population, and some undesirable complications due to the patients' existing comorbidities. Therefore, pain management strategies for patients undergoing hip surgery are based on a range of anesthesia techniques, including the use of opioids, neuraxial anesthesia (spinal, epidural, or a combination of them), nerve blocks, especially pericapsular nerve block (PENG), fascia iliaca compartment block (FICB) and femoral block). Reducing patients' pain and improving the quality of postoperative recovery has become increasingly important. The Quality of Recovery-15 (QoR-15) is a 15-question questionnaire validated to assess postoperative recovery. This questionnaire assesses patients' pain, physical comfort, physical independence, psychological support, and emotional status in the early postoperative period. The aim of this study was to evaluate the effect of ultrasound-guided PENG block, FICB block, and femoral block on the quality of recovery as part of multimodal analgesia before hip surgery under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* elective hip fracture,
* 18-85 years
* American Society of Anaesthesiology (ASA) I-III

Exclusion Criteria:

* patients planned for general anesthesia
* with multiple fractures
* bleeding disorder
* peripheral neuropathy
* mental disorder
* local anesthetic allergy
* contraindications for spinal anesthesia (local infection, etc.)
* declining to give written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include ASA I-III patients between the ages of 1-85 who are planned to undergo hip fracture surgery under elective spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-09-24 (Estimated); Study Completion 2024-10-24 (Estimated)

PRIMARY OUTCOMES:
recovery quality | 5 minutes
  The Quality of Recovery-15 (QoR-15) is a 15-question questionnaire validated to assess postoperative recovery. This questionnaire assesses patients' pain, physical comfort, physical independence, psychological support, and emotional status in the early postoperative period. The patient is asked to express their status scoring from 0 to 10; therefore, the total score ranges from 0 to 150 points,

SECONDARY OUTCOMES:
postoperative Numeric Rating Scale (NRS) pain score | postoperative 24 hours
  The postoperative pain intensity will be assessed with Numeric Rating Scale (NRS) scores (0 represents no pain and 10 represents the worst possible pain) at postoperative 24 hours.
postoperative opioid consumption | postoperative 24 hours
  The amount of postoperative opioid consumption will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, M.D., Principal Investigator — University of Health Sciences, Antalya Training and Research Hospital
Locations (1):
- University of Health Sciences, Antalya Training and Researh Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalashetty MB, Channappagoudar R, Alwandikar V, Naik DL, Hulakund SY, Guddad A. Comparison of Pericapsular Nerve Group Block with Fascia Iliaca Compartment Block in Adult Patients Undergoing Hip Surgeries: A Double-Blinded Randomized Control Study. Anesth Essays Res. 2022 Jul-Sep;16(3):397-401. doi: 10.4103/aer.aer_123_22. Epub 2022 Dec 9. PMID 36620112
- [Background] Kukreja P, Uppal V, Kofskey AM, Feinstein J, Northern T, Davis C, Morgan CJ, Kalagara H. Quality of recovery after pericapsular nerve group (PENG) block for primary total hip arthroplasty under spinal anaesthesia: a randomised controlled observer-blinded trial. Br J Anaesth. 2023 Jun;130(6):773-779. doi: 10.1016/j.bja.2023.02.017. Epub 2023 Mar 22. PMID 36964012